CLINICAL TRIAL: NCT02785367
Title: Changes of Gas Values in Cord Blood Versus Time and Temperature
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0042-46-tlv
Record Dates: First submitted 2016-05-25; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Abnormal; Birth
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cord blood samples (Experimental): 8 cord blood samples will be taken from the umbilical cord in 8 syringes of about 3 ml washed with Heparin.
  Interventions: Procedure: Cord blood samples

INTERVENTIONS:
Procedure: Cord blood samples — After delivery, 8 cord blood samples will be taken from the umbilical cord in 8 syringes of about 3 ml, washed with Heparin (Designated syringes exist in the delivery room). 4 syringes will be stored in room temperature. Thermometer will be attached to any sample, and temperature values will be indicated before any measurement.
  The samples will be measured in a gas measurement device, in 4 time points: at the birth, after 15 minutes, after 30 minutes and after 60 minutes from the birth.

SUMMARY:
The pH levels of a neonatal at his birth are an important factor in establishing the connection between events that occurred during the actual time of birth, to the risk of a significant morbidity development in the future. Gas values in cord blood are measurable and represent the condition of the fetus close to the time of birth. Their level is one of the essential criteria which are used to define acute hypoxic event during birth. As the oxygen supply to the fetus significantly disturbed, deficiency of oxygen in the tissues is growing. Therefore, the tissues begin to accumulate large amounts of acid and thereby developing fetal blood acidosis. Many works connected the presence of cord blood acidosis to development of neonatal cerebral palsy. According to the American Association of Obstetrics and Gynecology, cord blood gas sample is necessary when a prenatal event may be related (rightly or not) with negative neonatal outcome. This approach might be necessary when the case is legally controversial and there is a need to prove that umbilical cord gas values were normal at the prenatal period.

DETAILED DESCRIPTION:
The PH levels of a neonatal in his birth are an important factor in establishing the connection between events that occurred during the actual time of birth, to the risk of a significant morbidity development in the future. Gas values in cord blood are measurable and represent the condition of the fetus close to the time of birth. Their level is one of the essential criteria which are used to define acute hypoxic event during birth. As the oxygen supply to the fetus significantly disturbed, deficiency of oxygen in the tissues is growing. Therefore, the tissues begin to accumulate large amounts of acid and thereby developing fetal blood acidosis. Many works connected the presence of cord blood acidosis to development of neonatal cerebral palsy. According to the American Association of Obstetrics and Gynecology, cord blood gas sample is necessary when a prenatal event may be related (rightly or not) with negative neonatal outcome. This approach might be necessary when the case is legally controversial and there is a need to prove that umbilical cord gas values were normal at the pre-natal period.

Aim of study Our aim is to find the effect of the cord blood sample storage way, and the effect of the sample taking time from the delivery.

ELIGIBILITY:
Inclusion Criteria:

Gestational age 37 weeks and above. Vaginal or cesarean births.

Exclusion Criteria:

Women who had medical indication to cord blood sample taking for gas measurement (Apgar<7 in the 5th minute, premature labor (under 37 weeks), multiple pregnancy, vacuum birth, urgent cesarean

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
gas values | 60 minutes
  gas(pH) values will be examined at different times after the birth.

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No